CLINICAL TRIAL: NCT03669107
Title: Effect of Chewing Gum on Gastrointestinal Function Recovery After Surgery of Gynecological Cancer Patients at Rajavithi Hospital
Brief Title: Effect of Chewing Gum on Gastrointestinal Function Recovery After Surgery of Gynecological Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJchewinggum
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2018-10

CONDITIONS: Gum Chewing
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gum chewing (Experimental): Gum type was standardized with all subjects receiving sugar-free peppermint-flavored gum.
  The patients in the chewing gum group, gum chewing began the morning of postoperative day 1. Patients chewed gum (one stick) 3 times daily in the morning, afternoon, and evening at 30 min. The administration of the therapy was implemented by ward nursing staff and recorded in the patients file. All gum-chewing patients completed their course of gum chewing until bowel function.
  Interventions: Drug: Gum
- Control group (No Intervention): no gum

INTERVENTIONS:
Drug: Gum — no gum
  Arms: Gum chewing

SUMMARY:
A total patients undergoing abdominal complete surgical staging for various gynecological cancers were randomized into a gum-chewing group or a control group. The patients chewed sugarless gum three times from the first postoperative morning until the first passage of flatus. Each chewing session lasted 30 min. Total abdominal hysterectomy with systematic pelvic and para-aortic lymphad- enectomy was performed on all patients as part of complete staging surgery. Groups were compared in terms of time to first bowel movement time, first flatus and feces pass time, Total length of hospital stay.

DETAILED DESCRIPTION:
This study was conducted from September 2018-September, 2019 at Rajavithi Hospital, Department of Gynecologic Oncology.

Female patients preparing for complete surgical staging for malignant gynecologic disease such as endometrial cancer, cervix cancer and ovarian cancer were assessed for eligibility. Exclusion criteria for the study included thyroid diseases, inflammatory bowel disease, complaints of chronic constipation (defined as two or fewer bowel movements per week), a history of prior abdominal bowel surgery, abdominal radiation, or neoadjuvant chemotherapy, need for intensive care more that 24 h postoperatively, nasogastric tube drainage beyond the first postoperative morning, or bowel anastomosis and upper abdominal multivisceral surgical approaches in relation to the debulking surgery.

The study information was explained to all enrolled subjects, informed written consent obtained and randomization performed as soon as the patients were admitted to the investigator's gynecologic oncology service. Eligible patients were randomly assigned to one of two groups by an investigator (I.E.E.) by consecutive opening of sequentially numbered, opaque, sealed envelopes. Envelope randomization was performed by a blocked of four randomization method. Group A acted as the control group and received no treatment, and Group B received sugar-free peppermint-flavored chewing gum.

The same evidence-based protocol of perioperative management, except for chewing gum, was used for all patients. All patients underwent total abdominal hysterectomy with systematic pelvic and para- aortic lymph node dissection as part of their staging procedures. The same surgical team performed all operations.

All subjects received the same postoperative care regimen, All patients were mobilized as soon as possible in the postoperative period.

To reduce the effects of other variables, the postoperative feeding re- gime was standardized for the study patients: 30-60 ml of water and if tolerated other liquids were started from the first postoperative day until the first passage of flatus. Upon passing flatus, clear fluids and if tolerated semiliquid fiberless diet was allowed. Patients were allowed to progress to a solid diet according to the patient's toleration or the pas- sage of feces. Group B began chewing gum on postoperative day one and chewed gum three times daily. Each chewing lasted 30 min. The administration of therapy was implemented by nursing ward staff and recorded in the patients file. All gum-chewing patients completed their course of gum chewing until the return of bowel function.

ELIGIBILITY:
Inclusion Criteria:

* • Female patients preparing for complete surgical staging for malig- nant gynecologic disease such as endometrial cancer, cervix cancer and ovarian cancer were assessed for eligibility.
* age 18-60 yr
* good consciousness

Exclusion Criteria:

* Exclusion criteria for the study included thyroid diseases, inflammatory bowel disease, complaints of chronic constipation (defined as two or fewer bowel movements per week), a history of prior abdominal bowel surgery, abdominal radiation, or neoadjuvant chemotherapy, need for intensive care more that 24 h postoperatively, nasogastric tube drainage beyond the first postopera- tive morning, or bowel anastomosis and upper abdominal multivisceral surgical approaches in relation to the debulking surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
postoperative flatus pass time | an expected average of 48 hours
  The main outcome variable of the study was postoperative flatus pass time (hours from end of operation). Participants will be followed for the duration of the flatus pass time,

SECONDARY OUTCOMES:
duration of hospital stay | an expected average of 3 weeks ]
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

REFERENCES:
- [Result] Ertas IE, Gungorduk K, Ozdemir A, Solmaz U, Dogan A, Yildirim Y. Influence of gum chewing on postoperative bowel activity after complete staging surgery for gynecological malignancies: a randomized controlled trial. Gynecol Oncol. 2013 Oct;131(1):118-22. doi: 10.1016/j.ygyno.2013.07.098. Epub 2013 Jul 29. PMID 23906657